CLINICAL TRIAL: NCT03331692
Title: A Comparison of Efficacy of Clinical Parameters With Auditory Evoked Potentials in Monitoring of Adequate Course of General Anesthesia
Brief Title: Monitoring of Adequate Course of General Anesthesia
Acronym: MoDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Dariusz Tomaszewski, Adjunct professor, Military Institute od Medicine National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06101968-05
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Monitoring of Depth of Anesthesia; AAI Index
MeSH Terms: interventions — Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Intervention Model Description: Participants are assigned to intravenous or volatile anesthesia. In both groups both the clinical and instrumental monitoring of the proper level of anesthesia was analyzed.
Who Masked: Participant, Care Provider
Masking Description: During the anesthesia, in all the participants an AAI-A line ARX index was continuously monitored. The electrodes were placed after the induction of anesthesia.
  Intraoperatively, both auditory evoked potentials with AAI index and electroencephalogram with burst suppression analysis was recorded. Recorded data were blinded for anesthesiologists, so were not used for analysis of level of anesthesia during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA group (Other): The participants scheduled for elective ENT procedures or for elective discectomy. The surgery was performed under totally intravenous anesthesia.
  During procedure, monitoring of the proper level of general anesthesia both clinical and instrumental was performed.
  Interventions: Other: monitoring of the proper level of general anesthesia
- VA group (Other): The participants scheduled for elective ENT procedures or for elective discectomy. The surgery was performed under volatile anesthesia. During procedure, monitoring of the proper level of general anesthesia both clinical and instrumental was performed.
  Interventions: Other: monitoring of the proper level of general anesthesia

INTERVENTIONS:
Other: monitoring of the proper level of general anesthesia — The monitoring of the adequate level of general anesthesia was performed both clinically and instrumentally.
  Other Names: clinical monitoring; instrumental monitoring

SUMMARY:
Clinical monitoring is the most common method of adjustment of the appropriate level of general anesthesia. However, the episodes of intraoperative awareness are still reported, suggesting that clinical observations may not be sufficient in some cases. The objective of the study was to compare the efficacy of clinical and instrumental neuromonitoring with auditory evoked potentials in intraoperative analysis of the proper level of general anesthesia.

The patients scheduled for elective surgery were included into the study, and randomly divided into two groups. Patients in the first group (TIVA group) underwent intravenous, in the second group (VA group) underwent volatile anesthesia. The adequacy of anesthesia was analyzed with standard clinical parameters. All the participants were instrumentally monitored with AAI index. After the anesthesia patients received a questionnaire with the questions regarding possible intraoperative awareness.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for ENT procedures or discectomy,
* preoperative health status I or II according to ASA score.

Exclusion Criteria:

* patients below 18 or above 61 year old,
* ASA status III or higher,
* patients suffering from: (i) hearing problems or tinnitus, (ii) chronic inflammation of the ear, (iii) epilepsy, and (iv) mental disorders,
* pregnancy.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2012-04-20 (Actual); Primary Completion 2013-08-30 (Actual); Study Completion 2014-07-14 (Actual)

PRIMARY OUTCOMES:
Changes in AAI values in selected (16) time points. | T1: after premedication, just before the onset of anesthesia; T2: 30 seconds after intravenous administration of propofol; T3: just before the endotracheal intubation; T4: 60 seconds after the endotracheal intubation; T5: 5 minutes after the endotracheal

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Therapy, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saper CB, Chou TC, Scammell TE. The sleep switch: hypothalamic control of sleep and wakefulness. Trends Neurosci. 2001 Dec;24(12):726-31. doi: 10.1016/s0166-2236(00)02002-6. PMID 11718878
- [Background] Nelson LE, Guo TZ, Lu J, Saper CB, Franks NP, Maze M. The sedative component of anesthesia is mediated by GABA(A) receptors in an endogenous sleep pathway. Nat Neurosci. 2002 Oct;5(10):979-84. doi: 10.1038/nn913. PMID 12195434
- [Background] Lu J, Nelson LE, Franks N, Maze M, Chamberlin NL, Saper CB. Role of endogenous sleep-wake and analgesic systems in anesthesia. J Comp Neurol. 2008 Jun 1;508(4):648-62. doi: 10.1002/cne.21685. PMID 18383504
- [Background] Ghoneim MM, Block RI, Haffarnan M, Mathews MJ. Awareness during anesthesia: risk factors, causes and sequelae: a review of reported cases in the literature. Anesth Analg. 2009 Feb;108(2):527-35. doi: 10.1213/ane.0b013e318193c634. PMID 19151283
- [Background] Wang DS, Orser BA. Inhibition of learning and memory by general anesthetics. Can J Anaesth. 2011 Feb;58(2):167-77. doi: 10.1007/s12630-010-9428-8. Epub 2010 Dec 23. PMID 21181566
- [Background] Sebel PS, Bowdle TA, Ghoneim MM, Rampil IJ, Padilla RE, Gan TJ, Domino KB. The incidence of awareness during anesthesia: a multicenter United States study. Anesth Analg. 2004 Sep;99(3):833-839. doi: 10.1213/01.ANE.0000130261.90896.6C. PMID 15333419
- [Background] Osterman JE, Hopper J, Heran WJ, Keane TM, van der Kolk BA. Awareness under anesthesia and the development of posttraumatic stress disorder. Gen Hosp Psychiatry. 2001 Jul-Aug;23(4):198-204. doi: 10.1016/s0163-8343(01)00142-6. PMID 11543846